CLINICAL TRIAL: NCT01318317
Title: Phase I/II Study of Cellular Immunotherapy Using Central Memory-Enriched CD8+ T Cells Lentivirally Transduced to Express A CD19-Specific Chimeric Immunoreceptor Following Peripheral Blood Stem Cell Transplantation for Patients With High-Risk Intermediate Grade B-Lineage Non-Hodgkin Lymphoma
Brief Title: Genetically Engineered Lymphocyte Therapy After Peripheral Blood Stem Cell Transplant in Treating Patients With High-Risk, Intermediate-Grade, B-cell Non-Hodgkin Lymphoma
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09174; NCI-2011-00344 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09174 (Other: City of Hope Medical Center); P30CA033572 (NIH); P50CA107399 (NIH)
Record Dates: First submitted 2011-03-16; First posted 2011-03-18 (Estimated); Results first posted 2021-12-21 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Follicular; Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Stem Cell Transplantation; Filgrastim; Granulocyte Colony-Stimulating Factor; Peripheral Blood Stem Cell Transplantation; plerixafor; ferric pyrophosphate; Rituximab; CT-P10

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cellular adoptive immunotherapy following PBSCT) (Experimental): Patients receive standard salvage chemotherapy per standard practice and undergo standard mobilization for stem cell collection with G-CSF and/or plerixafor. Some patients may also receive rituximab IV within 4 weeks of transplant. Patients receive standard myeloablative conditioning followed by autologous PBSCT. Patients then undergo infusion of ex vivo expanded autologous TCM-enriched CD8+ T cells expressing CD19-specific CAR on day 2 or 3 after transplant.
  Interventions: Procedure: Autologous Hematopoietic Stem Cell Transplantation; Biological: Filgrastim; Biological: Genetically Engineered Lymphocyte Therapy; Other: Laboratory Biomarker Analysis; Procedure: Peripheral Blood Stem Cell Transplantation; Drug: Plerixafor; Biological: Rituximab

INTERVENTIONS:
Procedure: Autologous Hematopoietic Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: AHSCT; Autologous; Autologous Hematopoietic Cell Transplantation; Autologous Stem Cell Transplant; Autologous Stem Cell Transplantation; Stem Cell Transplantation, Autologous
Biological: Filgrastim — Given IV
  Other Names: Filgrastim-aafi; G-CSF; Neupogen; Nivestym; r-metHuG-CSF; Recombinant Methionyl Human Granulocyte Colony Stimulating Factor; rG-CSF; Tevagrastim
Biological: Genetically Engineered Lymphocyte Therapy — Receive ex vivo expanded autologous TCM-enriched CD8+ T cells expressing CD19-specific CAR
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Peripheral Blood Stem Cell Transplantation — Undergo autologous PBSCT
  Other Names: PBPC transplantation; PBSCT; Peripheral Blood Progenitor Cell Transplantation; PERIPHERAL BLOOD STEM CELL TRANSPLANT; Peripheral Stem Cell Support; Peripheral Stem Cell Transplant; Peripheral Stem Cell Transplantation
Drug: Plerixafor — Given IV
  Other Names: AMD 3100; JM-3100; Mozobil; SDZ SID 791
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab ABBS; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar JHL1101; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; Rituximab Biosimilar SIBP-02; rituximab biosimilar TQB2303; rituximab-abbs; RTXM83; Truxima

SUMMARY:
This phase I/II trial studies the side effects and best dose of genetically engineered lymphocyte therapy and to see how well it works after peripheral blood stem cell transplant (PBSCT) in treating patients with high-risk, intermediate-grade, B-cell non-Hodgkin lymphoma (NHL). Genetically engineered lymphocyte therapy may stimulate the immune system in different ways and stop cancer cells from growing. Giving rituximab together with chemotherapy before a PBSCT stops the growth of cancer cells by stopping them from dividing or killing them. Giving colony-stimulating factors, such as filgrastim (G-CSF), or plerixafor helps stem cells move from the bone marrow to the blood so they can be collected and stored. More chemotherapy or radiation therapy is given to prepare the bone marrow for the stem cell transplant. The stem cells are then returned to the patient to replace the blood-forming cells that were destroyed by the chemotherapy. Giving genetically engineered lymphocyte therapy after PBSCT may be an effective treatment for NHL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of cellular immunotherapy utilizing ex vivo expanded autologous central memory T cell (TCM)-enriched cluster of differentiation (CD)8+ T cells genetically-modified to express a CD19-specific chimeric antigen receptor (CAR) in conjunction with a standard myeloablative autologous hematopoietic stem cell transplantation (aHSCT) for research participants with high-risk intermediate grade B-lineage non-Hodgkin lymphomas who have relapsed after primary therapy, or who did not achieve complete remission with primary therapy. (Phase I) II. To determine the maximum tolerated dose (MTD) on dose limiting toxicities (DLTs) and to describe the full toxicity profile. (Phase I) III. To determine the rate of research participants receiving TCM-enriched CD8+ T cells genetically-modified to express a CD19-specific CAR for which the transferred cells are detected in the circulation 28 days (+/- 3 days) by woodchuck hepatitis virus post-transcriptional regulatory element (WPRE) quantitative (Q)-polymerase chain reaction (PCR). (Phase II)

SECONDARY OBJECTIVES:

I. To determine the tempo, magnitude, and duration of engraftment of the transferred T cell product as it relates to the number of cells infused. (Phase II) II. To study the impact of this therapeutic intervention on the development of CD19+ B-cell precursors in the bone marrow as a surrogate for the in vivo effector function of transferred CD19-specific T cells. (Phase II) III. To describe the progression-free and overall survival of treated research participants on this protocol. (Phase II)

OUTLINE: This is a phase I, dose-escalation study of genetically engineered lymphocyte therapy followed by a phase II study.

Patients receive standard salvage chemotherapy per standard practice and undergo standard mobilization for stem cell collection with filgrastim and/or plerixafor. Some patients may also receive rituximab intravenously (IV) within 4 weeks of transplant. Patients receive standard myeloablative conditioning followed by autologous PBSCT. Patients then undergo infusion of ex vivo expanded autologous TCM-enriched CD8+ T cells expressing CD19-specific CAR on day 2 or 3 after transplant.

After completion of study treatment, patients are followed up periodically for at least 15 years.

ELIGIBILITY:
Inclusion Criteria:

* City of Hope (COH) pathology review confirms that research participant's diagnostic material is consistent with history of intermediate grade B-cell NHL (e.g., diffuse B-cell lymphoma, mantle cell lymphoma, transformed follicular lymphoma)
* History of relapse after achieving first remission with primary therapy, or failure to achieve remission with primary therapy
* Life expectancy > 16 weeks
* Karnofsky performance scale (KPS) >= 70%
* Negative serum pregnancy test for women of childbearing potential
* Research participant has an indication to be considered for autologous stem cell transplantation

Exclusion Criteria:

* Fails to understand the basic elements of the protocol and/or the risks/benefits of participating in this phase I/II study; evidence of understanding includes passing the Protocol Comprehensive Screening given by the Research Subject Advocate (RSA); a legal guardian may substitute for the research participant
* Any standard contraindications to myeloablative HSCT per standard of care practices at COH
* Dependence on corticosteroids
* Currently enrolled in another investigational therapy protocol
* Human immunodeficiency virus (HIV) seropositive based on testing performed within 4 weeks of enrollment
* History of allogeneic HSCT or prior autologous HSCT
* Active autoimmune disease requiring systemic immunosuppressive therapy
* Research participant(s) who are to receive radioimmunotherapy (Zevalin-based)-based conditioning regimens
* Research participant(s) with known active hepatitis B or C infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2011-09-19 (Actual); Primary Completion 2013-10-03 (Actual); Study Completion 2026-02-26 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth L Budde, MD,PhD, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

REFERENCES:
- [Derived] Ernst M, Oeser A, Besiroglu B, Caro-Valenzuela J, Abd El Aziz M, Monsef I, Borchmann P, Estcourt LJ, Skoetz N, Goldkuhle M. Chimeric antigen receptor (CAR) T-cell therapy for people with relapsed or refractory diffuse large B-cell lymphoma. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD013365. doi: 10.1002/14651858.CD013365.pub2. PMID 34515338
- [Derived] Wang X, Popplewell LL, Wagner JR, Naranjo A, Blanchard MS, Mott MR, Norris AP, Wong CW, Urak RZ, Chang WC, Khaled SK, Siddiqi T, Budde LE, Xu J, Chang B, Gidwaney N, Thomas SH, Cooper LJ, Riddell SR, Brown CE, Jensen MC, Forman SJ. Phase 1 studies of central memory-derived CD19 CAR T-cell therapy following autologous HSCT in patients with B-cell NHL. Blood. 2016 Jun 16;127(24):2980-90. doi: 10.1182/blood-2015-12-686725. Epub 2016 Apr 26. PMID 27118452

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Three additional participants underwent leukapheresis, however, two were ineligible for transplant and the third refused additional treatment and therefore were not assigned a dose level.
Groups:
- Dose Level 0 (25 x 10^6 CAR+ T-cells); Dose Level 1 (50 x 10^6 CAR+ T-cells); Dose Level 2 (100 x 10^6 CAR+ T-cells): Patients receive standard salvage chemotherapy per standard practice and undergo standard mobilization for stem cell collection with Granulocyte-Colony Stimulating Factor (G-CSF) and/or plerixafor. All patients receive rituximab IV within 4 weeks of transplantation. Patients receive standard myeloablative conditioning followed by autologous Peripheral Blood Stem Cell Transplant (PBSCT). Patients then undergo infusion of ex vivo expanded autologous central memory (TCM)-enriched CD8+ T cells expressing CD19-specific chimeric antigen receptor (CAR) on day 2 or 3 after transplantation.
Period: Overall Study
Arm/Group | Dose Level 0 (25 x 10^6 CAR+ T-cells) | Dose Level 1 (50 x 10^6 CAR+ T-cells) | Dose Level 2 (100 x 10^6 CAR+ T-cells)
Started | 1 | 4 | 3
Completed | 1 | 4 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Dose Level 0 (25 x 10^6 CAR+ T-cells); Dose Level 1 (50 x 10^6 CAR+ T-cells); Dose Level 2 (100 x 10^6 CAR+ T-cells): Patients receive standard salvage chemotherapy per standard practice and undergo standard mobilization for stem cell collection with Granulocyte-Colony Stimulating Factor (G-CSF) and/or plerixafor. Some patients may also receive rituximab IV within 4 weeks of transplantation. Patients receive standard myeloablative conditioning followed by autologous Peripheral Blood Stem Cell Transplant (PBSCT). Patients then undergo infusion of ex vivo expanded autologous central memory (TCM)-enriched CD8+ T cells expressing CD19-specific chimeric antigen receptor (CAR) on day 2 or 3 after transplantation.
- Total: Total of all reporting groups
Arm/Group | Dose Level 0 (25 x 10^6 CAR+ T-cells) | Dose Level 1 (50 x 10^6 CAR+ T-cells) | Dose Level 2 (100 x 10^6 CAR+ T-cells) | Total
Number analyzed (Participants) | 1 | 4 | 3 | 8
Age, Continuous [Median (Full Range); unit: years] | 75 [NA to NA] — Only 1 participant in this dose level | 60 [50 to 69] | 58 [57 to 65] | 62 [50 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 1 | 4
  Male | 1 | 1 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 4 | 3 | 8
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 1 | 4 | 3 | 8
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 4 | 3 | 8
Disease histology [Count of Participants; unit: Participants]
  Diffuse Large B-Cell Lymphoma | 1 | 3 | 3 | 7
  Mantle Cell Lymphoma | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose Limiting Toxicities (DLTs)
Description: Number of DLTs per dose level are reported.
  A DLT is defined as:
  Any grade 3 or higher toxicity, with the exception of expected adverse events; and designated as definitely or probably related (level of attribution) to the infusion of the TCM cells; and occurring within 28 days of T-cell infusion; Any toxicity requiring the use of steroids to ablate side effects attributable to the infusion of the TCM cells, and occurring within 28 days of T-cell infusion; Any toxicity which is a lower grade, but that increases in grade to a grade 3 or higher as a direct result of the TCM, and occurring within 28 days of T-cell infusion; Any grade 2 or greater autoimmune toxicity, and occurring within 28 days of T-cell infusion.
Time Frame: Within 28 days of T-cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0 (25 x 10^6 CAR+ T-cells) | Dose Level 1 (50 x 10^6 CAR+ T-cells) | Dose Level 2 (100 x 10^6 CAR+ T-cells)
Number analyzed (Participants) | 1 | 4 | 3
Participants | 0 | 0 | 0

2. Primary Outcome: Woodchuck Hepatitis Virus Post-transcriptional Regulatory Element (WPRE) Detection Above Background
Description: Peak expansion of WPRE is expressed in CAR copy number/mL of blood is summarized with median and range
Time Frame: 28 days post T cell infusion
Population: 1 participant in dose level 1 did not have any whole blood samples to analyze. Overall median was reported due to small samples sizes in each dose level.
Measure: Median (Full Range); unit: CAR copy number/mL
Groups:
- Treatment (Cellular Adoptive Immunotherapy Following PBSCT): Patients receive standard salvage chemotherapy per standard practice and undergo standard mobilization for stem cell collection with Granulocyte-Colony Stimulating Factor (G-CSF) and/or plerixafor. Some patients may also receive rituximab IV within 4 weeks of transplantation. Patients receive standard myeloablative conditioning followed by autologous Peripheral Blood Stem Cell Transplant (PBSCT). Patients then undergo infusion of ex vivo expanded autologous central memory (TCM)-enriched CD8+ T cells expressing CD19-specific chimeric antigen receptor (CAR) on day 2 or 3 after transplantation.
  peripheral blood stem cell transplantation (PBSCT): Undergo autologous PBSCT
  filgrastim: Given IV
  polymerase chain reaction: Correlative studies
  rituximab: Given IV
  genetically engineered lymphocyte therapy: Receive ex vivo expanded autologous central memory (TCM)-enriched CD8+ T cells expressing CD19-specific chimeric antigen receptor (CAR)
  laboratory biomarker analysis: Correlative studies
  plerixafor: Given IV
  autologous hematopoietic stem cell transplantation: Undergo autologous PBSCT
Arm/Group | Treatment (Cellular Adoptive Immunotherapy Following PBSCT)
Number analyzed (Participants) | 7
CAR copy number/mL | 280 [0 to 925]

3. Primary Outcome: Number of Days of Quantifiable CD19 CAR Post T-cell Infusion
Description: WPRE persistence of quantifiable CD19 CAR summarized with mean and standard deviation
Time Frame: 28 days post T cell infusion
Population: 1 participant in dose level 1 did not have any whole blood samples to analyze. Overall mean was reported due to small samples sizes in each dose level.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Treatment (Cellular Adoptive Immunotherapy Following PBSCT)
Number analyzed (Participants) | 7
days | 18.25 (12.1)

4. Secondary Outcome: Failure to Engraft
Description: Count of participants who fail to engraft post transplant.
Time Frame: Within 21 days post T-cell infusion
Measure: Count of Participants; unit: Participants
Arm/Group | Dose Level 0 (25 x 10^6 CAR+ T-cells) | Dose Level 1 (50 x 10^6 CAR+ T-cells) | Dose Level 2 (100 x 10^6 CAR+ T-cells)
Number analyzed (Participants) | 1 | 4 | 3
Participants | 0 | 0 | 0

5. Secondary Outcome: Progression-free Survival at 1 Year
Description: Estimated using the Kaplan-Meier methods.
  Progression is defined using the revised IWG response criteria, as any new lesion or increase by ≥50% of previously involved sites from nadir.
Time Frame: Up to 1 year
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Cellular Adoptive Immunotherapy Following PBSCT)
Number analyzed (Participants) | 8
percentage of participants | 50 [16 to 84]

ADVERSE EVENTS:
Time Frame: During and after treatment, up to 38 months
Arm/Group | Dose Level 0 (25 x 10^6 CAR+ T-cells) | Dose Level 1 (50 x 10^6 CAR+ T-cells) | Dose Level 2 (100 x 10^6 CAR+ T-cells)
All-Cause Mortality (participants affected / at risk) | 0/1 | 1/4 | 1/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 2/4 | 3/3
Other Adverse Events (participants affected / at risk) | 1/1 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 0 (25 x 10^6 CAR+ T-cells) (N=1) | Dose Level 1 (50 x 10^6 CAR+ T-cells) (N=4) | Dose Level 2 (100 x 10^6 CAR+ T-cells) (N=3)
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0
Neoplasms benign, malignant, and unspecified (incl cysts and polyps)- Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Stroke (Nervous system disorders) | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 0 (25 x 10^6 CAR+ T-cells) (N=1) | Dose Level 1 (50 x 10^6 CAR+ T-cells) (N=4) | Dose Level 2 (100 x 10^6 CAR+ T-cells) (N=3)
Anemia (Blood and lymphatic system disorders) | 1 | 4 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 2 | 3
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 4 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 2
Constipation (Gastrointestinal disorders) | 1 | 2 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 4 | 3
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2
Fecal incontinence (Gastrointestinal disorders) | 0 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 2 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 3 | 2
Nausea (Gastrointestinal disorders) | 1 | 4 | 3
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Rectal pain (Gastrointestinal disorders) | 0 | 1 | 0
Rectal ulcer (Gastrointestinal disorders) | 0 | 0 | 1
Typhlitis (Gastrointestinal disorders) | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 3 | 3
Chills (General disorders) | 1 | 1 | 1
Fatigue (General disorders) | 1 | 4 | 3
Fever (General disorders) | 1 | 3 | 3
Injection site reaction (General disorders) | 0 | 1 | 0
Pain (General disorders) | 0 | 2 | 1
Edema limbs (General disorders) | 1 | 2 | 2
Infusion related reaction (General disorders) | 0 | 1 | 1
Localized edema (General disorders) | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 1 | 0
Catheter related infection (Infections and infestations) | 0 | 0 | 1
Eye infection (Infections and infestations) | 0 | 1 | 0
Infections and infestations - Other, specify (Infections and infestations) | 0 | 1 | 0
Upper respiratory infection (Infections and infestations) | 0 | 1 | 1
Soft tissue infection (Infections and infestations) | 1 | 0 | 0
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 0 | 0 | 1
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 2
Alkaline phosphatase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 3 | 3
Blood bilirubin increased (Investigations) | 0 | 0 | 1
Cholesterol high (Investigations) | 0 | 1 | 0
Creatinine increased (Investigations) | 0 | 3 | 3
Lymphocyte count decreased (Investigations) | 1 | 4 | 3
Lymphocyte count increased (Investigations) | 0 | 2 | 0
Neutrophil count decreased (Investigations) | 1 | 4 | 3
Platelet count decreased (Investigations) | 1 | 4 | 3
Weight loss (Investigations) | 0 | 2 | 3
White blood cell decreased (Investigations) | 1 | 4 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 4 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 1
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypernatremia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypertriglyceridemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 4 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 4 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 3 | 2
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3 | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 2 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 3 | 3
Paresthesia (Nervous system disorders) | 0 | 0 | 2
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1 | 1
Presyncope (Nervous system disorders) | 0 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 3 | 2
Confusion (Psychiatric disorders) | 0 | 2 | 0
Insomnia (Psychiatric disorders) | 1 | 2 | 2
Restlessness (Psychiatric disorders) | 1 | 2 | 1
Hematuria (Renal and urinary disorders) | 0 | 2 | 1
Proteinuria (Renal and urinary disorders) | 0 | 2 | 0
Renal colic (Renal and urinary disorders) | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Bladder spasm (Renal and urinary disorders) | 0 | 1 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1 | 1
Breast pain (Reproductive system and breast disorders) | 0 | 2 | 0
Testicular pain (Reproductive system and breast disorders) | 0 | 0 | 1
Vaginal pain (Reproductive system and breast disorders) | 0 | 1 | 0
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 3
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 3 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Erythema multiforme (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 3 | 2
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 4 | 3
Lymphedema (Vascular disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-10): https://cdn.clinicaltrials.gov/large-docs/17/NCT01318317/Prot_SAP_000.pdf